CLINICAL TRIAL: NCT05772962
Title: Children at Risk and Oral Health, The Dental Record Study
Status: Recruiting | Type: Observational
Sponsor: Oral Health Centre of Expertise in Western Norway (Other)
Collaborators: Childrens advocacy center Bergen Norway (Unknown); The public dental health service Vestland Norway (Unknown); Oral Health Center of Expertise Rogaland, Norway (Other)
Responsible Party: Sponsor
Other Study IDs: Children at risk
Record Dates: First submitted 2022-12-21; First posted 2023-03-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Child Abuse; Child Neglect; Child Maltreatment
Keywords: Oral health; Dental health service; Childrens advocacy center; Prevention; Detection; Collaboration

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children enrolled at CAC: Information regarding oral health will be gathered from the public dental health records of children enrolled at CAC.
- Children not enrolled at CAC: Information regarding oral health will be gathered from the public dental health records of children that have not been enrolled at CAC. This is a control group, matched by age and gender.

SUMMARY:
The objectives of this retrospective dental record study, are to increase knowledge of the oral health, - history and -needs of children enrolled at the Childrens Advocacy Centers (CAC)by:

* assessing if it is possible to identify oral indicators of child maltreatment.
* assessing if and to what degree the children enrolled at CAC are in need of close, adapted and trauma sensitive treatment and follow up at the Public Dental Health Service (PDHS)
* assessing if there is a need for new routines in terms of interdisciplinary collaboration and sharing of information between CAC, Child Welfare Services (CWS) and PDHP.

By increasing knowledge in regard to child maltreatment and oral health, the study will raise PDHS and CAC ability to prevent, detect and help children being victims of maltreatment, and contribute to strengthen PDHS, CAC and CWS interdisciplinary interaction for the benefit of children at risk.

DETAILED DESCRIPTION:
The combination of the CAC and the organization of the PDHS in Norway with regular summoning of all children up to 18 years, provides a unique opportunity to identify children at risk and study their oral health and history in a retrospective perspective. Retrospective dental record data will be collected from the public dental health records of children, aged 0-18 when enrolled at CAC, and a control group matched by gender and age.

In addition to increase knowledge of the oral health, and - history, the dental record data will also provide information regarding the PDHS 's ability to detect, follow up and interact with children at risk and to which degree interdisciplinary cooperation between the CAC, the child welfare service and the PDHS takes place and are functioning.

By using already existing data from the childrens dental records at the public dental health service the study will gain new and important knowledge, without adding further burden to the children and families.

The Ethical committee REK Vest, has approved the study and permitted that the study will be conducted without an informed consent from the parents and children being enrolled. In order to secure that the research project is in line with General Data Protection Regulation (GDPR), identify, evaluate and negating the risks of the personal data being collected, A Data Protection Impact Assessment (DPIA) has been conducted.

ELIGIBILITY:
Inclusion Criteria:

* Children enrolled at CAC
* Control group matched by age and gender

Exclusion Criteria:

* Children with developmental disorders that affect oral health
* Children with mental retardation

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children being between 0-18 years old at the time they are enrolled at CAC, and a matched controllgroup.
Sampling Method: Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2024-12-05 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Oral health and history | 2022-2024
  Assess if there are differences in oral health and history between children enrolled at CAC and the control group

SECONDARY OUTCOMES:
Need for facilitated dental treatment and follow up in the PDHS | 2022-2024
  Assess if and which needs children have is in regard to oral health, facilitated dental treatment in the PDHS, interdisciplinary collaboration and follow up. Are there differences between the two groups?

CONTACTS AND LOCATIONS:
Overall Officials: Ingfrid Vaksdal Brattabø, PhD, Principal Investigator — Oral Health Centre of Expertice, Western Norway
Locations (1):
- Oral Health Centre of Expertice Western Norway, Bergen, Vestland, Norway

IPD SHARING:
Plan to Share IPD: Undecided